CLINICAL TRIAL: NCT00803985
Title: A Randomised Controlled Trial Comparing Total Extra-Peritoneal (TEP) to Lichtenstein Inguinal Hernia Repair Concerning Physical Sequelae and Quality of Life at One and Three Years - the TEPLICH Trial
Brief Title: Study Comparing Total Extraperitoneal Patch "TEP" Versus Lichtenstein According Chronic Pain
Acronym: TEP-LICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Collaborators: Region Skane (Other)
Responsible Party: Principal Investigator, Agneta Montgomery, Assosiate professor, Skane University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 596/2007
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Chronic Pain; Sexual Dysfunction
Keywords: Inguinal hernia; TEP; Lichtenstein; Mesh; Randomized; Chronic pain; Sexual dysfunction
MeSH Terms: conditions — Chronic Pain; Sexual Dysfunction, Physiological; Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lichtenstein (Active Comparator): Open operation with onlay light weight polypropylene mesh
  Interventions: Procedure: Total Extraperitoneal repair (TEP)
- Total Extraperitoneal repair (TEP) (Active Comparator): Laparoscopic operation with preperitoneal nonfixated mesh
  Interventions: Procedure: Lichtenstein

INTERVENTIONS:
Procedure: Total Extraperitoneal repair (TEP) — Operation for primary inguinal hernias i men
  Other Names: Total extraperitoneal patch; Laparoscopic hernia operation; Hernia mesh operation
  Arms: Lichtenstein
Procedure: Lichtenstein — Operation for primary inguinal hernias i men
  Other Names: Open on lay mesh repair; Anterior mesh repair
  Arms: Total Extraperitoneal repair (TEP)

SUMMARY:
The purpose of this study is to se if there is a difference regarding chronic pain and sexual dysfunction one and tree years after laparoscopic un fixated preperitoneal mesh versus gold standard open fixated on lay mesh in inguinal hernia surgery.

Long term cross-sectional follow-up comparing different instruments for measurement of chronic pain.

DETAILED DESCRIPTION:
Prospective randomized study comparing total extraperitoneal patch TEP versus open onlay mesh according to Lichtenstein in primary unilateral inguinal hernias in men between 30 to 75 years of age. Non fixated polypropylene mesh is used in the TEP operation and fixated light weight polypropylene mesh is used in the Lichtenstein procedure. The aim is to study chronical pain and sexual dysfunction. Clinical examination according nerve function, hernia status and genital findings are performed together with a questionnaire including SF36, Inguinal Pain Questionnaire(IPQ), sexual function are registered preoperatively, one and tree years postoperatively.

Cross-sectional follow-up in median 7.5 years using enquiries for comparison of different pain instruments to evaluate the effect of chronic pain on physical activity.

ELIGIBILITY:
Inclusion Criteria:

* men between 30-75 years of age
* ASA class I-II
* primary unilateral inguinal hernia

Exclusion Criteria:

* lower midline incision below linea arcuate
* large scrotal hernia
* previously or current abuse,mental disease
* obesity BMI > 35
* another simultaneous operation
* nonreducible hernia
* severe pain in the groin without nonrelated to hernia
* contraindications to general anesthesia
* need of language translator
* liver cirrhosis or ascites
* spread cancer disease
* previously irradiation in the area
* lack of operations indication

Ages: 30 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Chronic pain during the last week (IPQ2) 1 year postoperatively measured using question 2 of the Inguinal Pain Questionnaire (IPQ). | One year
  The worst pain last week one year postoperatively. Measured using question 2 of IPQ-questionaire with the cutoff for pain set between grade 2 (pain present but could easily be ignored) and grade 3 (pain present but does not interfere with everyday activities)

SECONDARY OUTCOMES:
Quality of life measured using the SF-36 questionnaire | one and three years
  SF-36 is composed of eight sub-scales and the composite scores for physical and mental health. Norm-based scores were calculated using the Swedish age and gender specific means and standard deviations. The norm data have a mean of 50 and a standard deviation (SD) of 10. A 5-point difference corresponds to an effect size (Cohen's d) of 0.5 SD, which was regarded as a medium-sized clinical difference.
Chronic pain right now and during the last week (IPQ1 and IPQ2) measured using question 1 and 2 of the inguinal pain questionnaire. | IPQ1 grade 2-7, IPQ1 grade 3-7 and IPQ2 grade 2-7 measured at one and three years. IPQ2 grad 3-7 measured at three years.
  Chronic pain was measured using IPQ with the following cutoffs. "Any pain last week" (IPQ2 grade 2-7) and "any pain right now" (IPQ2 grade 2-7) at 1 and 3 years. "Pain right now" (IPQ1 grade 3-7) at 1 and 3 years and "pain last week" (IPQ2 grade 3-7) at 3 years
Clinical exam assessing groin complaints | Exams were performed preoperatively, at one and three years
  Clinical examination was performed assessing groin complaints were reported in six dimensions (no complaints, tenderness, decreased sensation to touch, decreased sensation to pricking, increased sensation to touch or pricking, radiation of pain) in five defined locations in the groin/scrotum area.
A newly developed SexIHS questionnaire designed to specifically address sexual dysfunction associated with a diagnosed inguinal hernia or following inguinal hernia surgery. | Mean 33 months after surgery
  The first 2 questions adressing whether the patient is sexually active and if they have pain during intercourse. The following questions address pain-related sexual dysfunction by describing pain frequency, pain intensity, erectile or ejaculatory dysfunction and symptoms of depression.
  Two additional questions aimed to describe localisation and type of pain. Scores in the questionnaire vary between 0-12.
Physical function score measuring the ability to perform common daily activities | The functional score was measured preoperatively, at one and three years
  Physical function was measured using a functional score that was created by assessing three daily activities. Climbing stairs, squatting and raising from bed Each activity was graded from 0-2 points (0 = no discomfort, 1 = mild/moderate discomfort, and 2 = severe discomfort in need of support) with a sum of all scores between 0-6.
Number of patients with a recurrence after TEP and Lichtenstein surgery | After one and three years
  Recurrence after TEP and Lichtenstein repair.
Number patients with a harmful event during surgery after TEP and Lichtenstein | After one and three years
  A harmful event was defined as an unplanned chronic inconvenient condition beyond therapy following surgery (e.g. testicular atrophy or pain that did not exist before operation).
Number of patients with a adverse events after TEP and Lichtenstein surgery | After one and three years
  An adverse event was defined as either a reoperation due to a postoperative complication within 3 years or severe pain defined as IPQ2 grade 5-7

CONTACTS AND LOCATIONS:
Overall Officials: Agneta Montgomery, MD, PhD, Principal Investigator — University of Lund
Locations (1):
- Regionala etikprövningsnämden i Lund, avd 2, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gutlic N, Gutlic A, Petersson U, Rogmark P, Montgomery A. Randomized clinical trial comparing total extraperitoneal with Lichtenstein inguinal hernia repair (TEPLICH trial). Br J Surg. 2019 Jun;106(7):845-855. doi: 10.1002/bjs.11230. PMID 31162663